CLINICAL TRIAL: NCT06290011
Title: A Clinical Study on the Efficacy of Cognitive Distraction Focus Relaxation Therapy Based on MR in the Treatment of Chronic Pain: a Multicenter, Randomized Controlled, Single Blind Clinical Study
Brief Title: A Clinical Study on the Efficacy of Cognitive Distraction Focus Relaxation Therapy Based on MR
Status: Recruiting | Type: Observational
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: XH-23-014
Record Dates: First submitted 2023-12-26; First posted 2024-03-04 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pain key group: mixed real pain treatment software, pain treatment scenarios in MR
  Interventions: Device: Pain key group
- Sham MR group: TV screen 2D treatment scene with the same content provided

INTERVENTIONS:
Device: Pain key group — mixed real pain treatment software, pain treatment scenarios in MR
  Groups: Pain key group

SUMMARY:
A prospective, single blind, randomized, parallel controlled trial was conducted to evaluate the analgesic effect and safety of MR based "cognitive distraction focus relaxation therapy" in patients clinically diagnosed with chronic moderate to severe pain

DETAILED DESCRIPTION:
Multi-center, prospective, single-blind, randomized and parallel controlled trials are used to evaluate the role and impact of "digital chronic pain treatment system equipment" based on MR mixed reality technology in the clinical basic treatment of patients clinically diagnosed with chronic pain.

ELIGIBILITY:
Inclusion Criteria:

1. 18-85 years old male and female;
2. Patients clinically diagnosed with chronic pain;
3. Chronic pain lasts for more than 3 months;
4. The average intensity of pain in the past month is 40mm and above (VAS);
5. Willing to abide by the relevant regulations of the experiment;

Exclusion Criteria:

1. Serious cognitive impairment;
2. Current or previous diagnosis of epilepsy, dementia, migraine or other neurological diseases may hinder the use of mixed reality or have adverse effects;
3. Symptoms of nausea or dizziness;
4. Sensitive to luminous screens;
5. No stereo vision or severe hearing impairment;
6. Eye, face or neck injuries, which hinder the comfortable use of glasses;
7. The evaluated patient GAD-7 questionnaire 10 points and above, PHQ-9 questionnaire 10 points or above;
8. Have used VR or MR and other related devices to treat pain;
9. Other clinical studies have been completed now or recently (the past 2 months);
10. Currently pregnant or planning to get pregnant during the study;
11. At present, or some immediate family members work in a digital health company or pharmaceutical company that provides acute and chronic pain treatment.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic pain lasts for more than 3 months;
Sampling Method: Probability Sample
Enrollment: 132 (Estimated)
Dates: Start 2023-10-11 (Actual); Primary Completion 2025-06-11 (Estimated); Study Completion 2025-06-11 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale/Score（VAS） | 3 days
  VAS pain score criteria ((0-10 points) 0 Points: painless; 3 points below: have a slight pain, can tolerate; 4 points- -6 points: patients with pain and affect sleep, and can still tolerate; 7 points-10 points: the patient has gradually intense pain, the pain is unbearable, affect appetite, affect sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Ke NA Ma, phd, Study Chair — studay chair
Locations (1):
- Ke Ma, Shanghai, Yangpu, China

IPD SHARING:
Plan to Share IPD: Undecided